CLINICAL TRIAL: NCT03746483
Title: A Phase 2, Open-Label, Multicenter, 2x2 Crossover Trial to Assess the Safety and Efficacy of MS1819-SD in Patients With Exocrine Pancreatic Insufficiency Due to Cystic Fibrosis
Brief Title: OPTION: A Trial to Assess the Safety & Efficacy of MS1819 in Patients With Exocrine Pancreatic Insufficiency Due to Cystic Fibrosis
Acronym: OPTION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Entero Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AZ-CF2001
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Results first posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2020-02

CONDITIONS: Exocrine Pancreatic Insufficiency (EPI); Cystic Fibrosis (CF)
Keywords: Exocrine pancreatic insufficiency; EPI; Cystic Fibrosis; CF; Pancreatic enzyme replacement therapy (PERT); Lipase
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: 2x2 Crossover
Masking Description: Unblinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MS1819 2240 mg/day (3 weeks) then PERT pre-study dose (3 weeks) (Experimental): Patients in arm will further be randomized to receive either the sequence consisting of MS1819 2240 mg/day for 3 weeks followed by PERT for another 3 weeks. During the PERT treatment period the patients will take their stable pre-study PERT dose.
  Interventions: Drug: MS1819; Drug: Porcine PERT
- PERT pre-study dose(3 weeks) then MS1819 2240 mg/day (3 weeks) (Experimental): Patients in arm will be randomized to receive PERT for 3 weeks followed by MS1819 2240 mg/day for another 3 weeks. During the PERT treatment period the patients will take their stable pre-study PERT dose.
  Interventions: Drug: MS1819; Drug: Porcine PERT

INTERVENTIONS:
Drug: MS1819 — MS1819, an oral, non-systemic, that is non-enterically-coated. It is a yeast-derived (non-porcine) lipase pancreatic enzyme replacement.
Drug: Porcine PERT — Porcine PERT is being used as a comparator to MS1819 as a second drug/intervention

SUMMARY:
The primary objectives of this study are to assess the safety and efficacy of MS1819-SD vs porcine pancreatic enzyme replacement therapy (PERT) in patients with exocrine pancreatic insufficiency (EPI) due to cystic fibrosis (CF).

DETAILED DESCRIPTION:
This is a Phase 2, open-label, multi-center, 2x2 crossover study assessing the safety and efficacy of MS1819-SD (spray dried) vs porcine PERT given at the same dose that was being administered during the pre-study period.

MS1819-SD will be assessed in a 2x2 crossover including at least 30 patients completing both periods.

ELIGIBILITY:
Inclusion Criteria:

1. Cystic fibrosis, based on 2 clinical features consistent with CF, plus initial diagnostic sweat chloride ≥ 60 mmol/L
2. Under stable dose of porcine PERT
3. A fair or better nutritional status
4. Fecal elastase <100 µg/g
5. Standard-of-care medications including Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) modulators are allowed

Exclusion Criteria:

1. History or diagnosis of fibrosing colonopathy
2. Any chronic diarrheal illness unrelated to pancreatic insufficiency
3. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥5 ×upper limit of normal (ULN), or total bilirubin level ≥1.5 ×ULN at the Screening visit
4. Feeding via an enteral tube during 6 months before screening
5. Forced expiratory volume ≤30% at the Screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-07-13 (Actual); Study Completion 2019-07-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (11):
  - Investigator Site 105, Long Beach, California
  - Investigator Site 102, Altamonte Springs, Florida
  - Investigator Site 107, Miami, Florida
  - Investigator Site 101, Glenview, Illinois
  - Investigator Site 111, Wichita, Kansas
  - Investigator Site 108, Portland, Maine
  - Investigator Site 103, Las Vegas, Nevada
  - Investigator Site 110, Cleveland, Ohio
  - Investigator Site 104, Toledo, Ohio
  - Investigator Site 106, Hershey, Pennsylvania
  - Investigator Site 109, Dallas, Texas
- Poland (3):
  - Investigator Site 203, Karpacz
  - Investigator Site 202, Rabka-Zdrój
  - Investigator Site 204, Sopot

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MS1819 2240 mg/Day (3 Weeks) Then PERT Pre-study Dose (3 Weeks): Participants were first randomized to receive MS1819 first and PERT during the crossover phase
- PERT Pre-study Dose (3 Weeks) Then MS1819 2240 mg/Day (3 Weeks): Participants were first randomized to receive PERT first and MS1819 during the crossover phase
Period: Overall Study
Arm/Group | MS1819 2240 mg/Day (3 Weeks) Then PERT Pre-study Dose (3 Weeks) | PERT Pre-study Dose (3 Weeks) Then MS1819 2240 mg/Day (3 Weeks)
Started | 21 | 20
Completed | 15 | 17
Not Completed | 6 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Population: modified intent-to-treat (mITT)
Groups:
- MS1819 - PERT Sequence: Participants were first randomized to receive MS1819 first and PERT during the crossover phase
- PERT - MS1819 Sequence: Participants were first randomized to receive PERT first and MS1819 during the crossover phase
- Total: Total of all reporting groups
Arm/Group | MS1819 - PERT Sequence | PERT - MS1819 Sequence | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 19 | 36
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (7.60) | 29.0 (7.97) | 28.8 (7.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 11 | 15
  Male | 13 | 8 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 19 | 35
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26
  Poland | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of MS1819-SD: Coefficient of Fat Absorption (CFA)
Description: The Coefficient of Fat Absorption (CFA%) is defined as:
  [72-hour fat intake (g) - 72-hour fat excretion (g)/72-hour fat intake(g)] x 100 = CFA% The threshold for CFA results (>80%) is considered clinically significant for treatment effectiveness by the FDA.
Time Frame: 3 weeks
Population: modified Intent To Treat (mITT)
Measure: Mean (Standard Deviation); unit: % CFA
Groups:
- MS1819: Measured while participants on MS1819
- PERT: Measured while participants on PERT
Arm/Group | MS1819 | PERT
Number analyzed (Participants) | 33 | 35
% CFA | 55.6 (21.44) | 86.2 (7.39)

2. Primary Outcome: Safety of MS1819-SD by Number of Participants Reporting 1 or More Adverse Events (AE)
Description: Number of participants reporting 1 or more adverse events
Time Frame: 6 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- MS1819: AE reported during treatment with MS1819
- PERT: AE reported during treatment with PERT
Arm/Group | MS1819 | PERT
Number analyzed (Participants) | 40 | 38
Participants
  Number of subjects with any TEAEs | 13 | 6
  Number of subjects with TEAEs related to | 2 | 0

3. Primary Outcome: Safety of MS1819-SD by Number of Treatment Emergent Adverse Events (TEAEs)
Description: Number of Treatment emergent adverse events
Time Frame: 6 weeks
Population: Safety Population
Measure: Number; unit: Number of TEAEs reported
Arm/Group | MS1819 | PERT
Number analyzed (Participants) | 40 | 38
Number of TEAEs reported
  Number of Treatment-emergent adverse event (TEAEs) | 19 | 8
  Number of serious TEAEs reported | 0 | 0

4. Secondary Outcome: Stool Weights
Description: The relative efficacy of MS1819-SD compared to porcine PERT will be assessed using stool weights
Time Frame: 6 weeks
Population: mITT. Samples from 4 patients were not available for analysis due to discontinuation from the study. Three patients discontinued in the MS1819 group while 1 patient discontinued in the PERT group.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | MS1819 | PERT
Number analyzed (Participants) | 33 | 35
grams | 1394.0 (590.63) | 727.3 (334.29)

5. Secondary Outcome: Signs and Symptoms of Malabsorption
Description: The relative efficacy of MS1819 compared to porcine PERT will be assessed using signs and symptoms of malabsorption. Abdominal pain, bloating, flatulence, increased stool quantity, and worsening of overall bowel habit were graded as 0 = none, 1 = mild, 2 = moderate, or 3 = severe.
Time Frame: 3 weeks
Population: Data presented at 3 weeks post first dose.
Measure: Count of Participants; unit: Participants
Arm/Group | MS1819 | PERT
Number analyzed (Participants) | 36 | 36
Participants
  Grade 0 | 15 | 32
  Grade 1 | 12 | 3
  Grade 2 | 6 | 1
  Grade 3 | 1 | 0
  Unknown | 2 | 0

6. Secondary Outcome: Coefficient of Nitrogen Absorption (CNA)
Description: CNA at the end of each treatment period was expressed as the percentage of nitrogen (protein) absorbed from the subjects diet.
Time Frame: 3 weeks per group.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: % CNA
Arm/Group | MS1819 | PERT
Number analyzed (Participants) | 33 | 35
% CNA | 93.0 (2.54) | 97.2 (1.21)

ADVERSE EVENTS:
Time Frame: ~11 weeks
Description: Number of participants reporting 1 or more adverse events (Affected)
Arm/Group | MS1819 | PERT
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/38
Other Adverse Events (participants affected / at risk) | 13/40 | 6/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MS1819 (N=40) | PERT (N=38)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2 (2) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Sinus Headache (Nervous system disorders) | 1 (1) | 0 (0)
Nephrolithiasia (Renal and urinary disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lower Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/83/NCT03746483/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT03746483/SAP_001.pdf